CLINICAL TRIAL: NCT02767206
Title: Evaluation of Gastroesophageal Varices in Cirrhotic and Non-cirrhotic Patients With Portal Hypertension by Transnasal Endoscopy.
Brief Title: Evaluation of Gastroesophageal Varices by Transnasal Endoscopy.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Anderson Antônio de Faria, Principal investigator Anderson Faria, Federal University of Minas Gerais
Other Study IDs: TransView
Record Dates: First submitted 2016-05-02; First posted 2016-05-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Esophageal Varices; Gastric Varices; Hypertension Portal; Liver Cirrhosis
Keywords: Transnasal endoscopy; ultrathin endoscopes; esophageal varices; gastric varices
MeSH Terms: conditions — Esophageal and Gastric Varices; Hypertension, Portal; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- portal hypertension: Patients with cirrhosis or non-cirrhotic portal hypertension.

SUMMARY:
The study aims to evaluate the feasibility of transnasal endoscopy in patients with portal hypertension, cirrhotic and non-cirrhotic. The incidence of the procedure's adverse effects, the patient's tolerance and his/her opinion about the exam are analyzed. In addition, the interobserver matched for the discoveries found in the study is carried out.

DETAILED DESCRIPTION:
It is a descriptive study that proposes to evaluate the feasibility of the transnasal endoscopy to screen for gastroesophageal varices in patients with portal hypertension, cirrhotic and non-cirrhotic. The rupture of gastroesophageal varices is the principal cause of death among cirrhotics, responsible for high rates of morbidity and mortality. Current medical literature recommends that the cirrhotic and the carriers of non-cirrhotic portal hypertension screen for gastric-esophageal varices in order to establish prophylactic and therapeutic measures, when recommended. Usually, the conventional peroral esophagogastroduodenoscopy is used for such purpose but the need for sedation reduces productivity, increases costs and introduces a small but not insignificant risk concerning complications, especially in decompensated cirrhotic. For this reason, a transnasal endoscopy would be an interesting option for these patients because it does not require sedation.

The patients will be referred to endoscopy unit from general hepatology and viral hepatitis ambulatory settings. All of those who were asked to undergo esophagogastroduodenoscopy to screen for gastroesophageal varices will be invited to participate in the study, as long as they fulfill the inclusion criteria and agree to participate and sign Consent Form.

After the endoscopy, a questionnaire will be filled out with information about the exam, tolerance, incidence of adverse effects and alterations that were found. This questionnaire will have information about the liver disease cause, the cirrhosis staging to evaluate the patient's disease gravity and the patient's perception of the exam. The endoscopy will register the alterations that were found and the data about the patient's monitoring. Besides, the alterations related to the portal hypertension and afterwards the images analyzed by another endoscopist will be photographed for the matched calculation.

The results will be submitted to analysis. Statistical differences will be calculated using test "t" of student or Chi-square and significant values (p) under 0.05 considered.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were age (older than 18), clinical, laboratory or histologic diagnosis of hepatic cirrhosis or portal hypertension, and agreement to participate in the study.

Exclusion Criteria:

* Refusal to submit to the procedure; refusal or inability to sign the term of consent; previous nasal surgery; coagulation disturbances considered as international normalized ratio more than 2, platelets below 40,000; current use of coumarins and heparin; history of repetition epistaxis; allergic rhinitis; nasal anatomic abnormality or known oropharynx; and infection of superior aerial ducts at the moment of the exam.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endoscopies were performed in patients between 18 and 70 years with clinical, laboratory or histologic cirrhosis. They included patients of both genders who had indicated to perform transnasal endoscopy for screening of gastroesophageal varices.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction through the visual analogue scale | immediate
  Patients will be interrogated about their perception related to transnasal EGD
Adverse events | immediate
  Patients will be monitored about adverse events related to the procedure

SECONDARY OUTCOMES:
interobserver agreement | 24 weeks
  endoscopic images will be assessed by different endoscopists to check for interobserver agreement

REFERENCES:
- [Background] Triantos C, Kalafateli M. Primary prevention of bleeding from esophageal varices in patients with liver cirrhosis. World J Hepatol. 2014 Jun 27;6(6):363-9. doi: 10.4254/wjh.v6.i6.363. PMID 25018847
- [Result] Aedo MR, Zavala-Gonzalez MA, Meixueiro-Daza A, Remes-Troche JM. Accuracy of transnasal endoscopy with a disposable esophagoscope compared to conventional endoscopy. World J Gastrointest Endosc. 2014 Apr 16;6(4):128-36. doi: 10.4253/wjge.v6.i4.128. PMID 24748920
- [Result] Ai ZL, Lan CH, Fan LL, Lan L, Cao Y, Li P, Song O, Chen DF. Unsedated transnasal upper gastrointestinal endoscopy has favorable diagnostic effectiveness, cardiopulmonary safety, and patient satisfaction compared with conventional or sedated endoscopy. Surg Endosc. 2012 Dec;26(12):3565-72. doi: 10.1007/s00464-012-2367-4. Epub 2012 Sep 14. PMID 22976847
- [Result] Alexandridis E, Inglis S, McAvoy NC, Falconer E, Graham C, Hayes PC, Plevris JN. Randomised clinical study: comparison of acceptability, patient tolerance, cardiac stress and endoscopic views in transnasal and transoral endoscopy under local anaesthetic. Aliment Pharmacol Ther. 2014 Sep;40(5):467-76. doi: 10.1111/apt.12866. Epub 2014 Jul 9. PMID 25039412
- [Result] Arantes V, Albuquerque W, Salles JM, Freitas Dias CA, Alberti LR, Kahaleh M, Ferrari TC, Coelho LG. Effectiveness of unsedated transnasal endoscopy with white-light, flexible spectral imaging color enhancement, and lugol staining for esophageal cancer screening in high-risk patients. J Clin Gastroenterol. 2013 Apr;47(4):314-21. doi: 10.1097/MCG.0b013e3182617fc1. PMID 23059405
- [Result] Assy N, Rosser BG, Grahame GR, Minuk GY. Risk of sedation for upper GI endoscopy exacerbating subclinical hepatic encephalopathy in patients with cirrhosis. Gastrointest Endosc. 1999 Jun;49(6):690-4. doi: 10.1016/s0016-5107(99)70283-x. PMID 10343210
- [Result] Atar M, Kadayifci A. Transnasal endoscopy: Technical considerations, advantages and limitations. World J Gastrointest Endosc. 2014 Feb 16;6(2):41-8. doi: 10.4253/wjge.v6.i2.41. PMID 24567791
- [Result] Bosch J, Pizcueta P, Feu F, Fernandez M, Garcia-Pagan JC. Pathophysiology of portal hypertension. Gastroenterol Clin North Am. 1992 Mar;21(1):1-14. PMID 1568769
- [Result] Boyer TD. Natural history of portal hypertension. Clin Liver Dis. 1997 May;1(1):31-44, x. doi: 10.1016/s1089-3261(05)70253-1. PMID 15562666
- [Result] Choe WH, Kim JH, Ko SY, Kwon SY, Kim BK, Rhee KH, Seo TH, Lee TY, Hong SN, Lee SY, Sung IK, Park HS, Shim CS. Comparison of transnasal small-caliber vs. peroral conventional esophagogastroduodenoscopy for evaluating varices in unsedated cirrhotic patients. Endoscopy. 2011 Aug;43(8):649-56. doi: 10.1055/s-0030-1256474. Epub 2011 Jun 9. PMID 21660907
- [Result] Ciriza de los Rios C, Fernandez Eroles AL, Garcia Menendez L, Carneros Martin JA, Diez Hernandez A, Delgado Gomez M. [Sedation in upper gastrointestinal endoscopy. Analysis of tolerance, complications and cost-effectiveness]. Gastroenterol Hepatol. 2005 Jan;28(1):2-9. doi: 10.1157/13070376. Spanish. PMID 15691461
- [Result] D'Amico G, Pagliaro L, Bosch J. Pharmacological treatment of portal hypertension: an evidence-based approach. Semin Liver Dis. 1999;19(4):475-505. doi: 10.1055/s-2007-1007133. PMID 10643630
- [Result] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356
- [Result] Graham DY, Smith JL. The course of patients after variceal hemorrhage. Gastroenterology. 1981 Apr;80(4):800-9. PMID 6970703
- [Result] Ilyas JA, Kanwal F. Primary prophylaxis of variceal bleeding. Gastroenterol Clin North Am. 2014 Dec;43(4):783-94. doi: 10.1016/j.gtc.2014.08.008. Epub 2014 Sep 22. PMID 25440925
- [Result] Jobe BA, Hunter JG, Chang EY, Kim CY, Eisen GM, Robinson JD, Diggs BS, O'Rourke RW, Rader AE, Schipper P, Sauer DA, Peters JH, Lieberman DA, Morris CD. Office-based unsedated small-caliber endoscopy is equivalent to conventional sedated endoscopy in screening and surveillance for Barrett's esophagus: a randomized and blinded comparison. Am J Gastroenterol. 2006 Dec;101(12):2693-703. doi: 10.1111/j.1572-0241.2006.00890.x. PMID 17227516
- [Result] Kawai T, Miyazaki I, Yagi K, Kataoka M, Kawakami K, Yamagishi T, Sofuni A, Itoi T, Moriyasu F, Osaka Y, Takagi Y, Aoki T. Comparison of the effects on cardiopulmonary function of ultrathin transnasal versus normal diameter transoral esophagogastroduodenoscopy in Japan. Hepatogastroenterology. 2007 Apr-May;54(75):770-4. PMID 17591059
- [Result] Lee SY, Kawai T. Transnasal route: new approach to endoscopy. Gut Liver. 2008 Dec;2(3):155-65. doi: 10.5009/gnl.2008.2.3.155. Epub 2008 Dec 31. PMID 20485641
- [Result] Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy; Lichtenstein DR, Jagannath S, Baron TH, Anderson MA, Banerjee S, Dominitz JA, Fanelli RD, Gan SI, Harrison ME, Ikenberry SO, Shen B, Stewart L, Khan K, Vargo JJ. Sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2008 Nov;68(5):815-26. doi: 10.1016/j.gie.2008.09.029. No abstract available. PMID 18984096
- [Result] Pungpapong S, Keaveny A, Raimondo M, Dickson R, Woodward T, Harnois D, Wallace M. Accuracy and interobserver agreement of small-caliber vs. conventional esophagogastroduodenoscopy for evaluating esophageal varices. Endoscopy. 2007 Aug;39(8):673-80. doi: 10.1055/s-2007-966351. Epub 2007 Jun 22. PMID 17583856
- [Result] ASGE Technology Committee; Rodriguez SA, Banerjee S, Desilets D, Diehl DL, Farraye FA, Kaul V, Kwon RS, Mamula P, Pedrosa MC, Varadarajulu S, Song LM, Tierney WM. Ultrathin endoscopes. Gastrointest Endosc. 2010 May;71(6):893-8. doi: 10.1016/j.gie.2010.01.022. No abstract available. PMID 20438882
- [Result] Stroppa I, Grasso E, Paoluzi OA, Razzini C, Tosti C, Andrei F, Biancone L, Palmieri G, Romeo F, Pallone F. Unsedated transnasal versus transoral sedated upper gastrointestinal endoscopy: a one-series prospective study on safety and patient acceptability. Dig Liver Dis. 2008 Sep;40(9):767-75. doi: 10.1016/j.dld.2008.02.033. Epub 2008 Apr 18. PMID 18424197
- [Result] Tao G, Xing-Hua L, Ai-Ming Y, Wei-Xun Z, Fang Y, Xi W, Li-Yin W, Chong-Mei L, Gui-Jun F, Hui-Jun S, Dong-Sheng W, Yue L, Xiao-Qing L, Jia-Ming Q. Enhanced magnifying endoscopy for differential diagnosis of superficial gastric lesions identified with white-light endoscopy. Gastric Cancer. 2014 Jan;17(1):122-9. doi: 10.1007/s10120-013-0250-1. Epub 2013 Mar 14. PMID 23494118
- [Result] Triantafillidis JK, Merikas E, Nikolakis D, Papalois AE. Sedation in gastrointestinal endoscopy: current issues. World J Gastroenterol. 2013 Jan 28;19(4):463-81. doi: 10.3748/wjg.v19.i4.463. PMID 23382625
- [Result] Trevisani L, Cifala V, Sartori S, Gilli G, Matarese G, Abbasciano V. Unsedated ultrathin upper endoscopy is better than conventional endoscopy in routine outpatient gastroenterology practice: a randomized trial. World J Gastroenterol. 2007 Feb 14;13(6):906-11. doi: 10.3748/wjg.v13.i6.906. PMID 17352021